CLINICAL TRIAL: NCT06459336
Title: Comparative Effects of Intensive and Distributed Constraint-induced Movement Therapy on Upper Extremity Function in Stroke Patients
Brief Title: Comparative Effects of Intensive and Distributed CIMT on Upper Extremity Function in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0279
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Stroke; upper extremity function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive constraint-induced movement therapy (Experimental): intensive protocol of CIMT of total 36 hours will be given in a week
  Interventions: Other: Intensive constraint-induced movement therapy
- Distributed constraint-induced movement therapy (Experimental): Distributed participants will total of 36 hours treatment for 8 weeks
  Interventions: Other: Distributed constraint-induced movement therapy

INTERVENTIONS:
Other: Intensive constraint-induced movement therapy — Intensive protocol of CIMT will be given for 6hrs for 6 days to make total of 36 hours
  Arms: Intensive constraint-induced movement therapy
Other: Distributed constraint-induced movement therapy — Distributed protocol of CIMT will be given for 2.25hrs two times a week for 8 weeks making total of 36 hours
  Arms: Distributed constraint-induced movement therapy

SUMMARY:
The main question this clinical trial is aims to answer is whether intensive and distributed constraint-induced movement therapy has similar effects on upper extremity function in participants with stroke. Participants will receive intensive protocol of CIMT for 6 hours for 6 days to make total of 36 hours while distributed protocol participants will receive 2.25 hours of training two times a week for 8 weeks making total of 36 hours.

DETAILED DESCRIPTION:
Many studies have examined the effects of constraint-induced movement therapy (CIMT) in upper extremity function in stroke patients. Literature has shown effectiveness of different CIMT protocols for stroke patients. Emerging research have demonstrated comparative efficacy of constraint-induced movement therapy with different physical therapy approaches i.e. bimanual intensive training, motor relearning programme for improving upper extremity function. But according to researcher's knowledge, the gap of current knowledge is that no study has directly investigated the comparative effectiveness of intensive and distributed CIMT in stroke patients and if intensive and distributed CIMT had similar motor outcomes in upper limb function after stroke

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* ischemic or hemorrhagic stroke
* Both genders eligible
* Gcs score ≥ 13
* Able to extend at least 10° at the fingers
* Able to extend at least 20° at the wrist
* Patients diagnosed with one side more affected(hemiplegia)
* Modified Ashworth scale score ≤2

Exclusion Criteria:

* severe, chronic systemic illness
* Epilepsy
* History of fall past 6 months
* Injections of botulinum toxin type A or operations on the UE within 6 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity | 8th week
  It is designed to assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. It consists of 30 items assessing motor function and 3 items assessing reflex function. The score most applicable to task performance is given from "0, inability," "1, beginning ability," to "2, normal" (total score range, 0-66).
Wolf motor function test | 8th week
  This test was designed to assess the motor ability of patients with moderate to severe upper extremity motor deficits in the laboratory and clinic. The original version of this test was developed by Dr. Steven L. Wolf, Emory University School of Medicine. The original version consisted of 21 items; the widely used version of the wolf motor function test consists of 17 items. it uses a Uses a 6-point ordinal scale i.e."0" means "does not attempt with the involved arm" to "5" means "arm does participate; movement appears to be normal."

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, Phd, Principal Investigator — Riphah International University
Locations (1):
- Hameed Latif Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang TN, Liang KJ, Liu YC, Shieh JY, Chen HL. Effects of Intensive Versus Distributed Constraint-Induced Movement Therapy for Children With Unilateral Cerebral Palsy: A Quasi-Randomized Trial. Neurorehabil Neural Repair. 2023 Feb-Mar;37(2-3):109-118. doi: 10.1177/15459683231162330. Epub 2023 Mar 28. PMID 36987387
- [Background] Kaneko T, Maeda M, Yokoyama H, Kai S, Obuchi K, Takase S, Horimoto T, Shimada R, Moriya T, Ohmae H, Amanai M, Okita Y, Takebayashi T. Therapeutic effect of adjuvant therapy added to constraint-induced movement therapy in patients with subacute to chronic stroke: a systematic review and meta-analysis. Disabil Rehabil. 2024 Sep;46(18):4098-4112. doi: 10.1080/09638288.2023.2269843. Epub 2023 Oct 19. PMID 37855247